CLINICAL TRIAL: NCT05862285
Title: An Open-Label, Multicenter Extension Study in Patients Previously Enrolled in a Genentech and/or F. Hoffmann-La Roche Ltd Sponsored Study
Brief Title: A Rollover Study for Participants Previously Enrolled in a Genentech and/or F. Hoffman-La Roche Sponsored Study
Acronym: UmbrellaMAX
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BX44273; 2022-003414-36 (EudraCT Number); 2023-504263-16-00 (EU CTIS Number)
Record Dates: First submitted 2023-05-01; First posted 2023-05-17 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — ipatasertib; Tiragolumab; atezolizumab; Bevacizumab; entrectinib; inavolisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Roche IMP(s) Monotherapy (Experimental): Participants will continue to receive Roche IMP(s) monotherapy as per parent protocol, until disease progression, loss of clinical benefit as judged by the investigator, death, withdrawal of study consent, unacceptable toxicity, pregnancy, participants non-compliance, if local access becomes available or study termination by the Sponsor, whichever occurs first.
  Interventions: Drug: Ipatasertib; Drug: Atezolizumab; Drug: Bevacizumab; Drug: Entrectinib; Drug: Inavolisib; Drug: Divarasib
- Roche Combined Agents (Experimental): Participants will continue to receive Roche IMP(s) in combination with other agent(s) as per parent protocol, until disease progression, loss of clinical benefit as judged by the investigator, death, withdrawal of study consent, unacceptable toxicity, pregnancy, participants non-compliance, if local access becomes available or study termination by the Sponsor, whichever occurs first.
  Interventions: Drug: Tiragolumab; Drug: Atezolizumab; Drug: Tiragolumab and Atezolizumab; Drug: Bevacizumab; Drug: Inavolisib; Drug: Divarasib

INTERVENTIONS:
Drug: Ipatasertib — Ipatasertib will be administered as a monotherapy at the same dose, schedule, and with the same administration guidelines that were in effect at the time of participants discontinuation from the parent study.
  Other Names: RO5532961
  Arms: Roche IMP(s) Monotherapy
Drug: Tiragolumab — Tiragolumab in combination with atezolizumab will be administered at the same dose, schedule, and with the same administration guidelines that were in effect at the time of participants discontinuation from the parent study.
  Other Names: RO7092284
  Arms: Roche Combined Agents
Drug: Atezolizumab — Atezolizumab will be administered as a monotherapy and in combination at the same dose, schedule, and with the same administration guidelines that were in effect at the time of participants' discontinuation from the parent study.
  Other Names: RO5541267
Drug: Tiragolumab and Atezolizumab — Tiragolumab and Atezolizumab in fixed dose combination administered intravenously (IV) at the same dose, schedule, and with the same administration guidelines that were in effect at the time of participants discontinuation from the parent study.
  Other Names: RO7538483
  Arms: Roche Combined Agents
Drug: Bevacizumab — Bevacizumab will be administered as a monotherapy or in combination with atezolizumab at the same dose, schedule, and with the same administration guidelines that were in effect at the time of participants discontinuation from the parent study.
  Other Names: RO4876646
Drug: Entrectinib — Entrectinib will be administered as a monotherapy at the same dose, schedule, and with the same administration guidelines that were in effect at the time of participants discontinuation from the parent study.
  Other Names: RO7102122
  Arms: Roche IMP(s) Monotherapy
Drug: Inavolisib — Inavolisib will be administered as a monotherapy or in combination at the same dose, schedule, and with the same administration guidelines that were in effect at the time of participants discontinuation from the parent study.
  Other Names: RO7113755
Drug: Divarasib — Divarasib will be administered as a monotherapy or in combination with atezolizumab or bevacizumab at the same dose, schedule, and with the same administration guidelines that were in effect at the time of participants discontinuation from the parent study.
  Other Names: RO7435846

SUMMARY:
The purpose of this extension study is to provide continued treatment with Roche investigational medicinal product (IMP[s]) monotherapy or Roche IMP(s) combined with other agent(s) or comparator agent(s) for eligible participants with cancer who are still on study treatment at the time of roll-over from the parent study and who do not have access to the study treatment locally.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for continuing Roche IMP-based therapy at the time of roll-over from the parent study, as per the parent study protocol OR
* Eligible for continuing the comparator agent(s) in a Genentech- or Roche-sponsored study as per the parent study protocol, with no access to commercially available comparator agent
* First dose of study treatment in this extension study will be received within 7 days of the treatment interruption window allowed by the parent study
* Continue to benefit from the Roche IMP-based therapy or comparator at the time of roll-over from the parent study as assessed by the investigator
* Ability to comply with the extension study protocol, per Investigator's judgement

Exclusion Criteria:

* Meet any of the study treatment discontinuation criteria specified in the parent study at the time of enrollment in this extension study
* Study treatment or comparator agent is commercially marketed in the participant's country for the participant-specific disease and is accessible to the participant
* Treatment with any anti-cancer treatment (other than treatment permitted in the parent study) during the time between last treatment in the parent study and the first dose of study treatment in this extension study
* Permanent discontinuation of all study treatment(s) or comparator agent(s) for any reason during the parent study or during the time between last treatment in the parent study and the first dose of study treatment in this extension study (if applicable)
* Ongoing SAE(s) that has not resolved to baseline level or Grade ≤1 from the parent study or during the time between the last treatment in the parent study and the first dose of study treatment in this extension study
* Concurrent participation in any therapeutic clinical trial (other than the parent study)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2033-03-01 (Estimated); Study Completion 2033-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Continued Access to Roche IMP(s)-Based Therapy and/or Comparator Agent(s) | Up to approximately 10 years
Number and Severity of Participants With Selected Adverse Events Assessed as per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 5.0 | Up to approximately 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (55):
- Belgium (3):
  - GHdC Site Les Viviers, Charleroi
  - AZ Groeninge, Kortrijk
  - UZ Leuven Gasthuisberg, Leuven
- Princess Margaret Cancer Center, Toronto, Ontario, Canada
- China (15):
  - Beijing Cancer Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - West China Hospital of Sichuan University, Chengdu
  - Sir Run Run Shaw Hospital, School of Medicine, Zhejiang University, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - The Second Affiliated Hospital of Anhui Medical University, Hefei
  - Meizhou People's Hospital, Meizhou
  - The 1st Affiliated Hospital of Nanchang Unversity, Nanchang
  - Jiangsu Province Hospital of Chinese Medicine, Nanjing
  - Fudan University Shanghai Cancer Center, Shanghai
  - Shanghai Geriatric Medical Center, Shanghai
  - First Affiliated Hospital of Medical College of Xi'an Jiaotong University, Xi'an
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang
  - Henan Cancer Hospital, Zhengzhou
- Costa Rica (2):
  - Clinica CIMCA, San José
  - ICIMED Instituto de Investigación en Ciencias Médicas, San José
- France (9):
  - Centre Francois Baclesse, Caen
  - Institut de Cancérologie de Bourgogne, Dijon
  - Hopital de la Timone, Marseille
  - Centre Régional de Lutte Contre Le Cancer Val D'aurelle Paul Lamarque, Montpellier
  - Institut de cancerologie du Gard, Nîmes
  - Hopital Tenon, Paris
  - ICO - Site René Gauducheau, Saint-Herblain
  - Institut Claudius Regaud, Toulouse
  - Gustave Roussy, Villejuif
- Greece (2):
  - General Hospital "G.Papanikolaou", Asvestochóri
  - Metropolitan General Hospital, Cholargós
- Japan (6):
  - Kyushu University Hospital, Fukuoka
  - Yokohama City University Medical Center, Kanagawa
  - Kanagawa Cancer Center, Kanagawa
  - National Cancer Center Hospital East, Kashiwa-shi
  - Saitama Cancer Center, Saitama
  - NHO Kinki-Chuo Chest Medical Center, Sakaishi
- Mexico (3):
  - Centro Medico Culiacan SA de CV, Culiacán, Sinaloa
  - Medical Care & Research, Mérida, Yucatán
  - Consultorio de Especialidad en Urologia Privado, Durango
- Russia (3):
  - Moscow City Oncology Hospital #62, Moscovskaya Oblast, Moscow Oblast
  - Russian Scientific Center of Roentgenoradiology, Moscow, Moscow Oblast
  - P.A. Herzen Oncological Inst., Moscow, Moscow Oblast
- South Korea (2):
  - Seoul National University Bundang Hospital, Seongnam-si
  - Asan Medical Center, Seoul
- Taiwan (4):
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital - Linkou, Taoyuan District
- Thailand (3):
  - Chulalongkorn Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Maharaj Nakorn Chiangmai Hospital, Chiang Mai
- United Kingdom (2):
  - Leicester Royal Infirmary, Leicester
  - Royal Marsden Hospital - Surrey, Surrey

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing